CLINICAL TRIAL: NCT00134810
Title: A Phase II Multicentre Multinational Prospective Randomised Double-blind Placebo-controlled Study Assessing the Efficacy and Safety of a Single Application of Three Doses of Dysport® in Patients With Upper Back Myofascial Pain Syndrome
Brief Title: Study to Assess the Efficacy and Safety of Dysport® in Upper Back Myofascial Pain Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-47-52120-722; 2004-001845-13 (EudraCT Number)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Myofascial Pain Syndromes
Keywords: Myofascial pain syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The main purpose of this study is to determine which is the best dose of a drug known as Dysport to give when treating one's type of upper back pain. The study will also examine the side effects of this treatment and its overall effect on one's disorder.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe pain in upper back
* Myofascial pain syndrome for more than 6 months
* Active trigger points in upper back

Exclusion Criteria:

* Fibromyalgia and other non-myofascial pain conditions of upper back
* Duration of myofascial pain syndrome no longer than 24 months
* Steroid injections during previous 3 months
* Anaesthetic injection at trigger points during previous 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05-18 (Actual); Study Completion 2006-05-18 (Actual)

PRIMARY OUTCOMES:
Change in pain score for 'overall pain of the day during activity' between baseline and Week 6

SECONDARY OUTCOMES:
Change in pain score for 'worst pain of the day during activity' between baseline and Week 6
Change in pain score for 'overall pain of the day at rest' between baseline and Week 6
Spontaneously reported adverse events and changes in physical examination and vital signs
Change in pain score for 'overall pain during activity' between baseline and Weeks 6, 12 and 16
Time to onset of pain relief
Change in each of the 8 dimensions of the Short Form Quality of Life questionnaire with 36 items (SF36) at Weeks 6, 12 and 16 from baseline
Change in the Hospital Anxiety and Depression Scale (HADS) anxiety score, depression score and aggregate score at Weeks 6, 12 and 16 from baseline
Clinical Global Impression of Change (CGIC) assessed using a 7-point numerical rating scale at Week 16
Patient's Global Impression of Change (PGIC) assessed using a 7-point numerical rating scale at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (22):
- Czechia (3):
  - Pain Treatment Centre, Anesthesiology & Resuscitation, St Ann Teaching Hospital, Brno
  - Dept Neurology, Teaching Hospital Olomouc, Olomouc
  - Institute of Rheumatology, Prague
- Germany (7):
  - Neurology Clinic, Klinikum der Ruhr-Universitat Bochum, Bochum
  - Schmerzzentrum Frankfurt, Frankfurt am Main
  - Schmerzzentrum Goppingen, Göppingen
  - Klinik fur Anaesthesiologie und Intensivtherapie, Jena
  - Neurologisch-Verhaltensmedizinische Schmerzklinik Kiel, Kiel
  - Clinic for Neurology, Westfalische Wilhelmsuniversitat, Münster
  - Aukammallee 33, Wiesbaden
- Italy (2):
  - Fondazione Salvatore Maugeri, Montescano
  - Azienda Ospedaliera di Padova, Padua
- Poland (4):
  - Centrum Kliniczno-Badawcze, Elblag
  - Osrodek Badan Klinicznych, Lublin
  - Nasz Lekarz NZOZ Praktyka Grupowa Lekarzy, Torun
  - Centrum Medyczne OSTEOMED NZOZ, Warsaw
- Hospital de Santa Maria, Lisbon, Portugal
- Spain (5):
  - Hospital Univ Germans Trias i Pujol, Badalona
  - Hospital de Traumatologia de la Vall d'Hebrón, Barcelona
  - Hospedale Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Morales Meseguer, Murcia